CLINICAL TRIAL: NCT01974570
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Study for the Assessment of Anti-hypertensive Effect and Safety of Marealis RPC (Refined Peptide Concentrate), in Healthy Subjects With Mild or Moderate Hypertension
Brief Title: Effect and Safety of Marealis RPC (Refined Peptide Concentrate) in Mild or Moderate Hypertensive Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Marealis AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13TBHM
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Prehypertension
Keywords: Prehypertension; Hypertension; Shrimp protein hydrolysate; Marine protein hydrolysate; Ambulatory blood pressure; Blood pressure
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marealis refined peptide concentrate (Experimental): Participants are provided in double blinded fashion to Marealis refined peptide concentrate
  Interventions: Dietary Supplement: Marealis refined peptide concentrate
- Placebo (Placebo Comparator): Participants are provided in double blinded fashion to Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Marealis refined peptide concentrate — 2 tablets, once per day before noon
  Arms: Marealis refined peptide concentrate
Dietary Supplement: Placebo — 2 tablets, once per day before noon
  Arms: Placebo

SUMMARY:
Hypertension is an important risk factor of cardiovascular (CVD) and renal diseases. Epidemiological studies show that there is a direct relationship between blood pressure and CVD, and cardiovascular mortality increases progressively throughout the range of blood pressure, including the prehypertensive range. There is also evidence from cell and animal studies that shrimp tissue hydrolysates may have higher ACE inhibitory activity than other marine protein hydrolysates. It is hypothesized that Marealis RPC (refined peptide concentrate)will lower systolic blood pressure in subjects with elevated blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 30 to 75 years inclusive (independent and home-living subject).
* If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation); OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result.
* Mild or moderate hypertension (SBP 140-160 mmHg and DBP ≤ 100mmHg) (mean of office blood pressure measurements at the two first study visits during run-in period (visits 1 (-4 week) and 2 (-2 week)). Average office SBP baseline to be as close to 150mm Hg (i.e. 147-149 mmHg) as possible.
* Body weight ≥60kg
* Stable body weight (self-reported weight gain or loss <5kg in the past three months)
* Has given voluntary, written, informed consent to participate in the study
* Agrees to comply with study procedures including willingness to fast at least 12 hours before blood samples and abstain from alcohol two days prior to blood sampling and blood pressure measurement and abstain from coffee at least 14 hours before blood pressure measurement and abstain from physical exercise at least 4 hours before blood pressure measurement

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Body mass index ≥ 35 kg/m2
* Antihypertensive drug treatment, regular high dose NSAID treatment, use of cyclosporine or tacrolimus
* Any history of cardiovascular disease (myocardial infarction, unstable angina pectoris, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, temporal ischemic attack) including stroke and congestive heart failure
* Dementia, hypertensive retinopathy, left ventricular dysfunction or peripheral artery disease
* Anemia, abnormal electrolytes, proteinuria, abnormal liver, kidney and thyroid function (except subjects on thyroid replacement therapy)
* Clinically significant laboratory results
* Any other clinically significant abnormality in hematology and/or biochemistry at the Investigator's discretion
* Secondary hypertension
* Diabetes (type 1 and type 2 diabetes)
* History of cancer or malignant disease within the past 5 years(excluding basal cell carcinoma)
* Any metabolic disease, gastrointestinal disorder or other clinically significant disease/disorder which in the Investigator's opinion could interfere with the results of the study or the safety of the subject
* Dietary restriction (fish and other seafood allergies, citrus allergies, multiple food allergies)
* Alcohol abuse and/or illicit drug consumption; subjects consuming more than 14 portions of alcohol per week (one portion = 1 oz. spirits or 4 oz. wine or 11oz. medium strength beer / cider) Smokers and tobacco/snuff/nicotine users
* Consumption of natural health products targeted to blood pressure lowering within 30 days before randomization and during the study
* Participation in a clinical research trial within 30 days prior to randomization or during the study
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in daytime ambulatory systolic blood pressure from baseline | 8 weeks
Change in office systolic blood pressure from baseline | 8 weeks

SECONDARY OUTCOMES:
Change in 24-hour and nighttime ambulatory systolic blood pressure from baseline | 8 weeks
Change in 24-hour, daytime and nighttime ambulatory diastolic blood pressure from baseline | 8 weeks
Changes in 24-hour, daytime and nighttime ambulatory systolic and ambulatory diastolic blood pressure from baseline | 4 weeks
Mean ambulatory systolic blood pressure (24-hour, daytime and nighttime) | Over 8 weeks
Mean ambulatory diastolic blood pressure (24-hour, daytime and nighttime) | Over 8 weeks
Change in office diastolic blood pressure from baseline | 8 weeks
Changes in office systolic and office diastolic blood pressure from baseline | 2 weeks
Changes in office systolic and office diastolic blood pressure from baseline | 4 weeks
Mean Office systolic blood pressure | Over 8 weeks
Mean Office diastolic blood pressure | Over 8 weeks

OTHER OUTCOMES:
Mean heart rate | Over 8 weeks
Mean fasting serum glucose | 8 weeks
Mean fasting serum lipids (total cholesterol, HDL-cholesterol, LDL-cholesterol, total triglycerides) | 8 weeks
Mean serum C-reactive protein | 8 weeks
Dietary variables from food records (energy, carbohydrates, fats, proteins, fiber and sodium) | Over 8 weeks
Mean urine sodium | 8 weeks
Biometrics: weight and BMI | 8 weeks
Blood safety parameters: complete blood count, electrolytes (Na, K, Cl), creatinine, eGFR, AST, ALT, GGT, bilirubin | 8 weeks
Adverse events | Over 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (13):
- Biofortis Inc., Addison, Illinois, United States
- Canada (10):
  - Dr. William O'Mahony Medicine Professional Corporation, Corunna, Ontario
  - Dr. Steven V. Zizzo Medicine Professional Corporation, Hamilton, Ontario
  - Milestone Research, London, Ontario
  - Schacter Medicine Professional Corporation, London, Ontario
  - KGK Synergize Inc., London, Ontario
  - Dr. Dorli Herman, London, Ontario
  - SKDS Research Inc., Newmarket, Ontario
  - Glencar Medical Inc., Sarnia, Ontario
  - Dr. Anil Gupta Medicine Professional Corporation, Toronto, Ontario
  - Devonshire Clinical Research, Woodstock, Ontario
- A-Pharma, s.r.o, Prague, Czechia
- Analyze and Realize GmBH Professional Group, Berlin, Germany

REFERENCES:
- [Derived] Musa-Veloso K, Paulionis L, Pelipyagina T, Evans M. A Randomized, Double-Blind, Placebo-Controlled, Multicentre Trial of the Effects of a Shrimp Protein Hydrolysate on Blood Pressure. Int J Hypertens. 2019 Aug 5;2019:2345042. doi: 10.1155/2019/2345042. eCollection 2019. PMID 31467699